CLINICAL TRIAL: NCT01743833
Title: Effects of Thoracic Orthopedic Manual Therapy and Biopsychosocial Variables on Signs of Shoulder Impingement: A Randomized Clinical Trial
Brief Title: Effects of Thoracic Orthopedic Manual Therapy and Biopsychosocial Variables on Signs of Shoulder Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: Texas Tech University (Other)
Responsible Party: Principal Investigator, Augustus Mazzocca, Director, New England Musculoskeletal Institute Chairman, Department of Orthopaedic Surgery, UConn Health
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: #11-135-3
Record Dates: First submitted 2012-11-30; First posted 2012-12-06 (Estimated); Last update posted 2017-04-26 (Actual); Status verified 2017-04

CONDITIONS: Shoulder Impingement
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Thoracic HVLAMT, Postive Message (Active Comparator): Thoracic HVLAMT with a positive message given prior to the intervention.
  Interventions: Other: Thoracic High Velocity, Low Amplitude Thrust Maneuver (HVLATM)
- Thoracic HVLATM, Neutral Message (Active Comparator): Thoracic HVLAMT with a neutral message given prior to the intervention.
  Interventions: Other: Thoracic High Velocity, Low Amplitude Thrust Maneuver (HVLATM)
- Scapular HVLATM, Positive Message (Active Comparator): Scapular HVLAMT with a positive message given prior to the intervention.
  Interventions: Other: Scapular High Velocity, Low Amplitude Thrust Maneuver
- Scapular HVLATM, Neutral Message (Active Comparator): Scapular HVLAMT with a neutral message given prior to the intervention.
  Interventions: Other: Scapular High Velocity, Low Amplitude Thrust Maneuver

INTERVENTIONS:
Other: Thoracic High Velocity, Low Amplitude Thrust Maneuver (HVLATM)
  Arms: Thoracic HVLAMT, Postive Message; Thoracic HVLATM, Neutral Message
Other: Scapular High Velocity, Low Amplitude Thrust Maneuver
  Arms: Scapular HVLATM, Neutral Message; Scapular HVLATM, Positive Message

SUMMARY:
Shoulder impingement has been identified as the most common cause of shoulder pain in the adult general population. Sometimes therapeutic pushing on the middle part of the back (manual therapy) decreases shoulder pain in someone experiencing shoulder impingement. We do not known what causes the decreased shoulder pain. It could be that the therapeutic pushing makes things move better. It may be that the person getting their back treatment thinks they are better or the physical therapist who provides the manual treatment thinks it works.

DETAILED DESCRIPTION:
Shoulder impingement has been identified as the most common cause of shoulder pain in the adult general population. High-Velocity, Low-Amplitude Thrust Manipulations (HVLATM) of the thoracic spine and ribs result in increased shoulder ROM, as well as decreased pain and disability in patients suffering shoulder impingement. The quality of the sparse publications is low and lacking control or comparison groups regarding the use of HVLATM in the management of shoulder impingement. Further higher quality randomized clinical trials are needed. Moreover, no research has investigated the effects of the patients beliefs and different types of verbal messages conveyed by the clinician to the subjects in regard to the effects of HVLATM of the thoracic spine on shoulder pain and function. The purpose of this study is to evaluate, in subjects with signs and symptoms of shoulder impingement: (1) the effects of a series of the prone thoracic spine High Velocity Low Amplitude Thrust Manipulation (HVLATM) as compared to the HVLATM directed at the scapula, on shoulder pain, impingement symptoms, and functional outcomes; (2) the effect of the type of message and language used by the clinician in regard to thoracic HVLATM on shoulder pain, impingement symptoms, and functional outcomes; (3) the effect of subject's expectation of outcome of thoracic and scapula HVLATM on shoulder pain, impingement symptoms, and functional outcomes; (4) if these potential immediate improvements will be sustained at 6 to 9-day follow up.

ELIGIBILITY:
Inclusion Criteria:

* A consecutive convenience sampling of patients with complaints of shoulder pain that are not post-surgical will be screened at their initial evaluation. Subjects between the ages of 18 and 69 years will be included if they present with a painful arc of shoulder active ROM. Additional requirements for inclusion will be (1) shoulder pain greater than 1/10 but less than 9/10 at time of testing; (2) shoulder active ROM above horizontal; (3) the ability to lie prone with arms at their side; and (4) at least one of the following signs or symptoms: (1) a positive Hawkins-Kennedy Sign; (2) a positive Neer Impingement Sign; (3) painful resisted abduction; (4) painful resisted external rotation at 0°of abduction with the elbows bent to 90°

Exclusion Criteria:

* Subjects will be excluded from the study if they have any of the following: (1) A history of unstable thoracic spine joints or fractures; (2) A history of spinal bone tumors; (3) A bleeding disorder or the use of anticoagulant therapy (not to include a baby aspirin); (4) Acute rheumatoid arthritis or ankylosing spondylitis; (5) Signs and symptoms of myelopathy or cauda equina syndrome; (6) A systemic infection that may involve the spinal column, ribs, or shoulder girdle; (7) A history of osteoporosis or fracture of shoulder girdle bones; (8) Presence of radiculopathy with progressive signs; (9) Primary complaints of neck or thoracic pain; (10) A positive cervical distraction test; (11) A positive Spurling's test; (12) A large three-dimensional limitation of arm motion of greater than 20 degrees with any passive motion of the shoulder as compared to the contralateral side, to rule out adhesive capsulitis.; (13) A previous history of shoulder surgery such as a rotator cuff repair; (14) Physical therapy treatment to the shoulder or thoracic spine within the 3 months prior to participation in the study; (15) A cortisone or other fluid injection into the shoulder joint within 30 days of participation in the study; (16) A history of multiple sclerosis, or neuropathy; (17) Pregnancy; (18) Inability to attend a 6 to 9-day follow-up; and (19) Spinal fusion.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2011-06; Primary Completion 2012-12-05 (Actual); Study Completion 2012-12-05 (Actual)

PRIMARY OUTCOMES:
Shoulder Pain and Disability Index (SPADI) | 6-9 days following treatment
  The primary outcome measure is SPADI score at 6-9 days post intervention. The SPADI is also collected pretreatment and immediately post treatment.

SECONDARY OUTCOMES:
Numeric Pain Rating Scale | Pre, Post, and 6-9 days following treatment

OTHER OUTCOMES:
5 point Likert scale to asses effects of messaging (positive vs. neutral) | Pre-intervention

CONTACTS AND LOCATIONS:
Locations (1):
- University of Connecicut Health Center, Farmington, Connecticut, United States

REFERENCES:
- [Derived] Riley SP, Cote MP, Swanson B, Tafuto V, Sizer PS, Brismee JM. The Shoulder Pain and Disability Index: Is it sensitive and responsive to immediate change? Man Ther. 2015 Jun;20(3):494-8. doi: 10.1016/j.math.2014.12.002. Epub 2014 Dec 20. PMID 25560477
- [Derived] Riley SP, Bialosky J, Cote MP, Swanson BT, Tafuto V, Sizer PS, Brismee JM. Thoracic spinal manipulation for musculoskeletal shoulder pain: Can an instructional set change patient expectation and outcome? Man Ther. 2015 Jun;20(3):469-74. doi: 10.1016/j.math.2014.11.011. Epub 2014 Dec 2. PMID 25543999